CLINICAL TRIAL: NCT00741520
Title: Cardiovascular Impact of Obstructive Sleep Apnea in Normotensive Patients and the Effects of Continuous Positive Airway Pressure
Brief Title: Cardiovascular Impact of Obstructive Sleep Apnea Treatment in Normotensive Patients
Acronym: OSA-NORMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Geraldo Lorenzi-Filho, Heart Institute (InCor)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2431/04/051
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2008-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Blood Pressure; PreHypertension; Masked Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Prehypertension; Masked Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Control group
  Interventions: Device: CPAP
- 2 (Active Comparator): CPAP
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Control - no treatment
  Arms: 1
Device: CPAP — CPAP: The airway pressure will be determined by an overnight sleep study titration.
  Arms: 2

SUMMARY:
Recent evidences suggest that obstructive sleep apnea (OSA) can contribute to cardiovascular disease even in the absence of hypertension. However, there are few data regarding the impact of OSA on the preHypertension and Masked Hypertension in apparently normotensive patients with OSA as well as the impact of treatment with continuous positive airway pressure.

ELIGIBILITY:
Inclusion Criteria:

* Severe OSA patients

Exclusion Criteria:

* Smoking
* Sustained Hypertension
* Heart failure
* Diabetes
* Renal diseases
* Under use of any medication
* Under treatment for OSA

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Office Blood Pressure
  Evaluation of PreHypertension

SECONDARY OUTCOMES:
24 Hour Ambulatory Blood Pressure Monitoring
  Evaluation of Masked Hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor), São Paulo, São Paulo, Brazil